CLINICAL TRIAL: NCT03945006
Title: An Investigation of Balance, Trunk Impairment, and Fear of Falling in Multiple Sclerosis Patients With Incontinence
Brief Title: Balance, Trunk Impairment and Fear of Falling in Multiple Sclerosis Patients With Incontinence
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 72
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-03

CONDITIONS: Multiple Sclerosis; Physical Therapy; Incontinence
Keywords: Multiple Sclerosis; Balance; Trunk impairment; Fear of falling; Incontinence
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple Sclerosis Patients with Incontinence: Multiple Sclerosis with incontinence 24-58 years of age and being volunteered.
  Interventions: Other: Incontinence Severity; Other: Balance; Other: Trunk impairment; Other: Fear of falling
- Multiple Sclerosis Patients without incontinence: Multiple Sclerosis without incontinence 24-58 years of age and being volunteered.
  Interventions: Other: Incontinence Severity; Other: Balance; Other: Trunk impairment; Other: Fear of falling

INTERVENTIONS:
Other: Incontinence Severity — The Incontinence Severity Index (ISI) was used to assess the MS patients' incontinence severity.The first item is scored between 1 and 4 and the second item is scored between 1 and 3. The total score is calculated by the multiplication of these two answers. The index score is classified as 1-2 slight, 3-6 moderate, 8-9 severe, and 12 very severe.
  Other Names: Evaluation
Other: Balance — The patients were assessed while their bladders were empty. The static balance of the patients was measured with a Technobody® stabilometric platform. The patients were assessed while their bladders were empty. The test was performed as the patients' arms on the sides, eyes open and closed, and on two feet. Ellipse area, anterior-posterior sway, and medial-lateral sway scores were recorded.
  Other Names: Evaluation
Other: Trunk impairment — Trunk impairment was assessed with the Trunk Impairment Scale (TIS) while the participants' bladders were empty. The scale evaluates static and dynamic sitting balance and trunk coordination through 17 items. Each item is scored between 0 and 3. The total score ranges between 0 and 23, and higher scores indicate a better balance performance.
  Other Names: Evaluation
Other: Fear of falling — Fear of falling was assessed using the Falls Efficacy Scale developed by Tinetti and colleagues. The scale has 10 items assessing the effect of fear of falling on the confidence level of the individuals while performing activities of daily living. Each items is scored by the participants between 0 (not at all concerned) and 10 (very concerned), and the total of the score ranges between 0 (low fall efficacy) and 100 (high fall efficacy)
  Other Names: Evaluation

SUMMARY:
The aim of the present study was to examine balance, trunk impairment, and fear of falling in MS patients with incontinence. Clinical symptoms of the MS patients are heterogenous, and they vary according to the lesion levels and the duration and the type of the disease. In the neurologic group,especially in MS patients, incontinence is observed even at early stages.

Pelvic floor muscles contribute to continence by stabilizing the bladder neck and increasing the intraurethral pressure. Furthermore, they mechanically support the spine and the pelvis.This mechanical support is attained through an increase in sacroiliac joint stiffness and intra-abdominal pressure changes, which are important for spinal control. Along with incontinence, this mechanical support deteriorates resulting in some problems. By this way, postural function of pelvic floor muscles may alter in individuals with incontinence, and thus, lumbopelvic stabilization may be negatively affected. In addition, the activity of trunk muscles changes in individuals with incontinence, which may result in spinal movement and affect the posture. Therefore, balance disorders may develop. Postural sways caused by balance disorders and the decrease in postural corrections have been listed among risk the factors associated with falling.

When literature is examined, there exists no study examining the effects of incontinence on balance, trunk impairment, and fear of falling in MS patients. For all these reasons, investigators think that incontinence in MS patients has an effect on balance, trunk impairment, and fear of fall.

DETAILED DESCRIPTION:
This study was aimed to investigate balance, trunk impairment, and fear of falling in MS patients with and without incontinence.

The study was conducted in 35 MS patients with an age range of 24-58 years. The patients were divided into two groups based on the occurrence of incontinence. A neurologic examination was performed using the EDSS by a neurologist.

Incontinence was measured with the Incontinence Severity Index (ISI), balance was measured with a Technobody® stabilometric platform, and fear of falling was measured with the Falls Efficacy Scale (FES).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Multiple Sclerosis Disease
* The level of disability should be between 0.5-4 according to EDSS
* having a score of 24 or more in the Mini Mental Status Test

Exclusion Criteria:

* Patients with acute attacks (six months prior to the study)
* Mini-Mental State Examination (MMSE) score of less tahn 25 points
* History of shoulder injury, surgery, medical problems or other neurological disorders in any of the participants

Ages: 24 Years to 58 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: multiple sclerosis with incontinence and multiple sclerosis without incontinence
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Assessment of the Severity of Incontinence | 3 week
  The Incontinence Severity Index (ISI) was used to assess the MS patients' incontinence severity. The first item is scored between 1 and 4 and the second item is scored between 1 and 3. The total score is calculated by the multiplication of these two answers. The index score is classified as 1-2 slight, 3-6 moderate, 8-9 severe, and 12 very severe.

SECONDARY OUTCOMES:
Static Balance Assessment | 3 week
  The static balance of the patients was measured with a Technobody® stabilometric platform. The test was performed as the patients' arms on the sides, eyes open and closed, and on two feet. Ellipse area, anterior-posterior sway, and medial-lateral sway scores were recorded. As the sway increases, the balance disorder increases.
Trunk Impairment Assesment | 3 week
  Trunk impairment was assessed with the Trunk Impairment Scale. The scale evaluates static and dynamic sitting balance and trunk coordination through 17 items. Each item is scored between 0 and 3. The total score ranges between 0 and 23, and higher scores indicate a better balance performance.
Fear of Falling | 3 week
  Fear of falling was assessed using the Falls Efficacy Scale. The scale has 10 items assessing the effect of fear of falling on the confidence level of the individuals while performing activities of daily living. Each items is scored by the participants between 0 (not at all concerned) and 10 (very concerned), and the total of the score ranges between 0 (low fall efficacy) and 100 (high fall efficacy).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences,Department of Physiotherapy and Rehabilitation, Ankara, Esenboğa, Turkey (Türkiye)